CLINICAL TRIAL: NCT01121887
Title: Motivational Interviewing in Smoking Cessation: A Controlled Clinical Trial at the Swedish National Tobacco Quitline
Brief Title: Telephone-based Treatment for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Asgeir R. Helgason & Lars Forsberg, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAN046684 / LS04010116; CAF2006-ASG (Other Grant/Funding Number: Cancerfonden)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2008-09

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; telephone counselling; motivational interviewing; treatment integrity; Tobacco Smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment (Active Comparator)
  Interventions: Behavioral: Standard treatment
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Standard treatment — Telephone-based smoking cessation counselling based on a combination of coaching and cognitive behavioural therapy (CBT) techniques. Counsellors are also trained in giving tailored advice regarding the use of smoking cessation aids.
  Clients are offered a choice between "reactive treatment" (clients initiate all contact) and "proactive treatment" (counsellors call back at appointed dates). Printed information material tailored to clients' needs is offered free of charge.
  Arms: Standard treatment
Behavioral: Motivational Interviewing — Telephone-based smoking cessation counselling with Motivational Interviewing added to the standard treatment protocol.
  Clients are offered a choice between "reactive treatment" (clients initiate all contact) and "proactive treatment" (counsellors call back at appointed dates). Printed information material tailored to clients' needs is offered free of charge.
  Arms: Motivational Interviewing

SUMMARY:
Aim: to assess the effect of adding Motivational Interviewing (MI) to the existing smoking cessation treatment protocol at the Swedish National Tobacco Quitline (SNTQ).

Methods: Experienced counsellors at SNTQ either received further training in the standard treatment (ST) protocol (including Cognitive Behavioural Therapy (CBT)) or a comprehensive regime of training in MI. 1309 clients were randomized to either the ST group or the group with MI added to the treatment protocol. In order to ensure treatment integrity among counsellors, MI skill was assessed using the Motivational Interviewing Treatment Integrity Code (MITI).

ELIGIBILITY:
Inclusion Criteria:

* Clients have to express a desire for support regarding smoking cessation
* Clients have to be willing to confirm their identity by answering a baseline registration questionnaire

Exclusion Criteria:

* Clients with obvious difficulties understanding Swedish
* Clients with obvious mental impairments
* Clients using tobacco products other than cigarettes (mainly smokeless tobacco, or "snus")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1309 (Actual)
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence | 12 months after initial contact with SNTQ
  Not one puff of smoke during the previous 7 days

SECONDARY OUTCOMES:
Continuous abstinence | 12 months after initial contact with SNTQ
  Not a single puff of smoke within the past six months or more

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir R Helgason, PhD, Principal Investigator — Karolinska Institutet; Lars Forsberg, PhD, Study Director — Karolinska Institutet
Locations (1):
- Asgeir R. Helgason, Stockholm, Sweden

REFERENCES:
- [Background] Helgason AR, Tomson T, Lund KE, Galanti R, Ahnve S, Gilljam H. Factors related to abstinence in a telephone helpline for smoking cessation. Eur J Public Health. 2004 Sep;14(3):306-10. doi: 10.1093/eurpub/14.3.306. PMID 15369039
- [Background] Nohlert E, Tegelberg A, Tillgren P, Johansson P, Rosenblad A, Helgason AR. Comparison of a high and a low intensity smoking cessation intervention in a dentistry setting in Sweden: a randomized trial. BMC Public Health. 2009 Apr 30;9:121. doi: 10.1186/1471-2458-9-121. PMID 19405969
- [Result] Forsberg L, Berman AH, Kallmen H, Hermansson U, Helgason AR. A test of the validity of the motivational interviewing treatment integrity code. Cogn Behav Ther. 2008;37(3):183-91. doi: 10.1080/16506070802091171. PMID 18608316
- [Result] Forsberg L, Kallmen H, Hermansson U, Berman AH, Helgason AR. Coding counsellor behaviour in motivational interviewing sessions: inter-rater reliability for the Swedish Motivational Interviewing Treatment Integrity Code (MITI). Cogn Behav Ther. 2007;36(3):162-9. doi: 10.1080/16506070701339887. PMID 17852172
- See also: Karolinska Institutet — http://www.ki.se